CLINICAL TRIAL: NCT06667739
Title: A Behaviour Change Intervention Promoting Physical Activity Following Dysvascular Amputation: a Pilot Study
Brief Title: Promoting Physical Activity Following Dysvascular Amputation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-001-WP
Record Dates: First submitted 2024-08-23; First posted 2024-10-31 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Amputation; Lower Limb Amputation Knee
Keywords: Physical activity; Behaviour change; Peer coaching
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This pilot study is a parallel group randomized controlled trial with an embedded qualitative component.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, masking to receipt (or not) of the intervention is impossible. One assessor will collect all data. They will be masked to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IMPACT-L3 (Experimental): The experimental group will receive virtual peer health coaching (~30 minutes weekly) delivered by a peer trainer over 8 weeks. Peer trainers with dysvascular LLA themselves will be matched to a participant based on gender and level of amputation. The peer will help participants set goals and create an action plan for physical activity. Peers will receive specialized training in brief action planning. Participants will have access to five web-based modules. Modules include content on benefits of physical activity, types of physical activity (strengthening, aerobic, balance, flexibility), intensity of activity (light, moderate, vigorous), and exercise safety. Participants will complete modules weekly at their own pace for the first 5 weeks. To support behaviour change, participants will be provided with a wearable to track their physical activity: an Apple Watch to be worn at the wrist of the non-dominant side.
  Interventions: Behavioral: IMPACT-L3
- Control (No Intervention): The control group will continue with their usual health care and be offered the intervention program at the end of the follow-up period (wait-list control).

INTERVENTIONS:
Behavioral: IMPACT-L3 — The intervention is a physical activity behaviour change intervention: IMproving Physical Activity through Coaching and Technology following Lower Limb Loss (IMPACT-L3). Two theories provide a framework for IMPACT-L3. One is social cognitive theory and the other is self-determination theory. As mHealth solutions have the potential to increase access and improve health outcomes, IMPACT-L3 will be delivered entirely virtually.
  Arms: IMPACT-L3

SUMMARY:
Loss of a lower limb due to diabetes can have a devastating impact on physical and mental health and quality of life. Individuals are at risk of other diseases such as cardiovascular disease, loss of the other limb and death. Physical activity can reduce risk of chronic disease and improve health outcomes; however, physical activity levels in people with limb loss are low, often due to reduced balance and walking ability. Rehabilitation services are not readily available and the cost of delivering such programs remains high. Working with individuals with lower limb amputation, we created a virtual, peer-led physical activity behaviour change intervention called IMproving Physical Activity through Coaching and Technology following Lower Limb Loss (IMPACT-L3). We will conduct a pilot study to assess feasibility and optimize design of a future trial of effectiveness.

DETAILED DESCRIPTION:
Background and Importance: Diabetes-related lower limb amputation (LLA) is a leading cause of disability globally, impacting individuals' physical and mental health and ultimately their quality of life. Individuals with LLA due to diabetes or other vascular disease (dysvascular LLA) often have comorbidities, including higher rates of cardiovascular disease than the general population. They are at risk of amputation in the contralateral limb and have high mortality rates (30% at one year).

There is strong evidence demonstrating that physical activity reduces risk of chronic disease and mortality and improves quality of life. However, people with dysvascular LLA often have reduced strength, balance, walking ability and increased energy expenditure during ambulation. Consequently, they have impaired mobility that can lead to sedentary behaviour. Across studies examining physical activity in people with dysvascular LLA, step counts ranged from 1250 steps/day in older prosthesis users to 3809±2189 steps/day in people with diabetes-related LLA. Unfortunately, limited availability of rehabilitation services for people with LLA and the high cost of delivering healthcare interventions makes provision of support for physical activity challenging. To address this gap, we co-created a physical activity intervention, IMproving Physical Activity through Coaching and Technology following Lower Limb Loss (IMPACT-L3), to support physical activity behaviour change in people with dysvascular LLA. Prior to launching a large trial, a pilot study is required to assess feasibility and optimize design of a future trial. This study aims to assess the feasibility of conducting a definitive randomized controlled trial (RCT) to determine the effectiveness of a virtual peer-led physical activity intervention on levels of physical activity and self-efficacy in people with dysvascular LLA. Specific objectives are to: 1) evaluate feasibility according to indicators of process, resources, management and treatment; 2) explore perceptions of program characteristics, program implementation and study procedures among individuals with LLA; 3) explore the perceived feasibility and acceptability of the program among peer coaches; and 4) inform a sample size calculation for a future trial of effectiveness.

Methods: This pilot study is a parallel group RCT with an embedded qualitative component. The intervention group will have access to once-weekly virtual peer coaching sessions with a gender and level of amputation-matched peer trained in brief action planning; web-based physical activity modules; and a wearable activity monitor for 8 weeks. The control group will continue their usual health care and be offered the intervention at the end of the follow-up period. Data on feasibility of implementing the intervention and conducting the trial will be collected including assessment of process, resource, management and treatment indicators. Progression Criteria: A traffic light approach (red, amber, green) will be used to guide the research team in determining what changes may be required to address identified challenges based on the indicators and in determining the feasibility of progression to a trial. The proposed primary outcomes for a future trial will be measured at baseline, post intervention (week 9) and 4 week follow-up: total physical activity counts per day measured by the ActiGraphTM activity monitor and self-efficacy measured by the Self-efficacy for Exercise scale. Other outcome measures include: the Physical Activity Scale for Individuals with Physical Disability, Frenchay Activity Index, the Center for Epidemiologic Studies Depression Scale, Activities-specific Balance Confidence scale, Prosthesis Evaluation Questionnaire - Mobility Section, and Short Form Health Survey 12 Item survey. Semi-structured interviews will explore feasibility and acceptability of the intervention to participants (~15-20 participants) and peers. Inductive thematic analysis will be employed to analyze qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* Dysvascular LLA (LLA due to diabetes or vascular disease)
* major LLA (at the ankle or above)
* living in the community
* adult at least 18 years of age
* comfortable communicating in English and able to understand basic English
* receptive to using a phone or tablet (e.g., to enable peer coaching, access to modules.

Exclusion Criteria:

* actively receiving rehabilitation services related to physical activity/mobility
* recommended medical supervision for physical activity by health care provider, or skin problems preventing usual activity
* not able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Consent rate: the percent of recruited individuals who provide consent per month. | 8 weeks
Withdrawal Rate: the percent of study participants withdrawing by 9 weeks and 4 week follow-up | enrollment to 13 weeks
Peer coach adherence: total number of peer coaching sessions attended by the peer-trainer. | enrollment to 8 weeks
Participant and tester burden: the amount of time it took to administer study outcomes at T1, T2, and T3 and the acceptability of the evaluation time commitment from the perspective of participants. | Baseline, end of intervention (week 9) and 4 week follow-up
Feasibility of data collection: percentage of participants with complete data on each measure at each evaluation time point. | Baseline, end of intervention (week 9) and 4 week follow-up
  For accelerometers, the percentage of devices that were returned at baseline and follow-up.
Participant processing time: time from initial contact to enrollment. | 8 weeks
Intervention fidelity: study-specific checklist outlining key components of the intervention completed by peers. | enrollment to 8 weeks
  A subset of peer coaching sessions will be recorded and reviewed by research staff.
Adverse events: the number of adverse events that occurred during physical activity for the intervention. | enrollment to 8 weeks
  Adverse events (e.g., falls) will be documented by peers on the standardized form used at each coaching sessions.
Usage of web-based module: number of completed modules and number of logins. | enrollment to 8 weeks
Participant recruitment rate: the number and proportion of participants recruited per month | 8 weeks
Peer recruitment: number of peers recruited | 2 years
Participant adherence: the percentage of peer coaching sessions participants attend. | enrollment to 8 weeks
The theoretical framework of acceptability (TFA) questionnaire | week 9
  Description: A brief questionnaire developed to assess acceptability in the design, evaluation and implementation of interventions.

SECONDARY OUTCOMES:
Objective physical activity | Baseline, week 9, 4 week follow-up
  A tri-axial accelerometer is a lightweight device used to measure total activity counts. The sum of the total count for the day will be used and averaged over the measurement period.
Self-efficacy for Exercise Scale | Baseline, week 9, 4 week follow-up
  A self-report measure (9 items) that includes situations that may influence physical activity participation. Participants will respond to each item on a 0 (not very confident) to 10 (very confident) scale.
Self-Regulatory Efficacy for Exercise | Baseline, week 9, 4 week follow-up
  8-item measure to assess participants' confidence in their ability to manage their exercise.
Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline, week 9, 4 week follow-up
  The CES-D will assess participant&amp;amp;amp;amp;amp;amp;#39;s self-rated depressive symptoms. It is a 20-item scale that refers to symptoms in the last week.
The Physical Activity Scale for Individuals with Physical Disability (PASIPD) | Baseline, week 9, 4 week follow-up
  The PASIPD is a 13-item questionnaire with subscales measuring leisure time, household and work-related activities.
Leisure-Time Physical Activity for People with Disabilities Questionnaire (LTPAQ-D) | Baseline, week 9, 4 week follow-up
  The LTPAQ-D is a self-report measure that assesses minutes of mild-, moderate-, and vigorous-intensity leisure time physical activity (i.e., activity that requires physical exertion and that one chooses to do in their free time performed over the past 7 days.
Activities-specific Balance Confidence scale (ABC) | Baseline, week 9, 4 week follow-up
  ABC is a self-report measure used to assess perceived balance confidence.
Prosthesis Evaluation Questionnaire - Mobility Section (PEQ-MS) | Baseline, week 9, 4 week follow-up
  The PEQ-MS score will be used to measure the amount of difficulty completing locomotion tasks.
Short Form Health Survey 12 Item survey (SF-12) | Baseline, week 9, 4 week follow-up
  The SF-12 will be used to measure health related quality of life.
Frenchay Activities Index (FAI) | Baseline, week 9, 4 week follow-up
  The 15-item FAI captures information on social activities. The items reflect the frequency of performance of basic and instrumental activities of daily living over three domains.
Self Efficacy for Exercise: Dysvascular Lower Limb Amputees | Baseline, week 9, 4 week follow-up
  4-item measure will be administered in addition the standardized self-efficacy for exercise measure and self-regulatory efficacy for exercise measure to address contextual factors relevant to dysvascular lower limb amputees.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal MacKay, PhD, Principal Investigator — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No